CLINICAL TRIAL: NCT01123915
Title: A Phase 1, Dose Escalating, Single Centre, Double Blind Study of the Safety and Immunogenicity of Opal-HIV-Gag Clade C in HIV Positive Subjects
Brief Title: A Safety and Immunogenicity Study of 3 Doses of Opal Immunotherapy in HIV Infected People
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Collaborators: Phillip T. and Susan M. Ragon Foundation (Unknown); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Opal-HIV-1001; 2008-005142-23 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2011-11

CONDITIONS: HIV Infections
Keywords: HIV; Therapeutic; Immunotherapy; Acquired Immunodeficiency Syndrome; Virus Diseases; Lentivirus Infections; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Virus Diseases; Lentivirus Infections | interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opal-HIV-Gag(c) (Experimental): Opal-HIV-Gag(c) administered ex vivo to separated white blood cells on 4 occasions at 4 weekly intervals.
  Interventions: Biological: Opal-HIV-Gag(c) Low Dose; Biological: Opal-HIV-Gag(c) Medium dose; Biological: Opal-HIV-Gag(c) High dose
- Diluent (Placebo Comparator): Administered ex vivo to separated white blood cells on 4 occasions at 4 weekly intervals.
  Interventions: Other: Dimethyl Sulfoxide

INTERVENTIONS:
Biological: Opal-HIV-Gag(c) Low Dose
  Arms: Opal-HIV-Gag(c)
Biological: Opal-HIV-Gag(c) Medium dose
  Arms: Opal-HIV-Gag(c)
Biological: Opal-HIV-Gag(c) High dose
  Arms: Opal-HIV-Gag(c)
Other: Dimethyl Sulfoxide
  Arms: Diluent

SUMMARY:
This phase I study is the first step to determine if Opal immunotherapy may have potential utility as a treatment for HIV. Although effective treatments for HIV infection exist, they are limited by the requirement for life-long daily treatment, cost, side effects, and the development of resistance.

There is a need for therapeutic approaches that induce or enhance T-cell immunity to control HIV disease. Overlapping Peptide-pulsed Autologous Cells (Opal) is a technique where autologous peripheral blood mononuclear cells (PBMC) or whole blood is pulsed with sets of overlapping peptides spanning whole proteins of HIV.

DETAILED DESCRIPTION:
Opal-HIV-Gag(c) is not for direct injection and is administered by ex vivo incubation of whole blood or separated blood components (such as white blood cells or peripheral blood mononuclear cells) and reinfusion.

As a practical alternative to PBMC separation and to optimise vaccine presentation during the ex vivo incubation, a blood cell separation device will be used to separate the whole blood and enrich the white blood cell component. The device processes whole blood in a closed, single use disposable kit. Reconstituted Opal-HIV-Gag(c)or matching placebo will be added to the white blood cells, incubated for one hour and reinfused into the subject. Subjects will receive 4 administrations at 4 weekly intervals. Subjects are followed for 12 weeks after the final administration.

Each dose group will be enrolled sequentially, with a sentinel group for each dose group. Satisfactory safety data from each cohort, reviewed by a Data Safety Monitoring Board, will permit dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Documented laboratory diagnosis of HIV 1 infection
* Documented HIV clade of infection
* 18 - 60 years of age, inclusive
* Stable antiretroviral therapy (ART) regimen containing at least 3 active ART agents for at least 2 months prior to Baseline
* Plasma HIV-Ribonucelc acid (RNA) <400 copies/millilitre (mL) for 6 months up to and including Screening. Subjects on stable ART with a single value ≥400 copies/mL (i.e. the result is unconfirmed by subsequent testing) within this timeframe may be included at the discretion of the Investigator
* CD4+ T-cell count ≥350 cells/cubic millimetres (mm3) at Screening (with nadir ≥100 cells/mm3)
* A positive immunogenic response when stimulated with HIV-1 Gag clade C peptides at Screening
* Male or female. Women of child-bearing potential must be using two effective methods of contraception and agree to continue to do so from Screening, throughout study medication dosing and for 28 days after the last dose of study medication

Exclusion Criteria:

* Any serious or active medical or psychiatric illness which, in the opinion of the Investigator, would interfere with treatment, assessment, compliance with the protocol, or subject safety. This would include any active clinically significant renal, cardiac, pulmonary, vascular, or metabolic (thyroid disorders, adrenal disease) illness, or malignancy
* Hepatitis B virus surface antigen, or Hepatitis C virus (HCV) antibody and HCV-RNA positive at Screening
* Female subjects who are lactating and those of reproductive potential with a positive urine pregnancy test at either Screening or Baseline
* A new AIDS-defining condition diagnosed within 42 days prior to Baseline visit
* Known or suspected allergy to Dimethyl Sulfoxide
* History of allergy or reaction to medications (including peptide or protein containing agents) or history of severe allergy that, in the opinion of the Investigator, might compromise the subject's participation in any way
* Moderate or severe asthma, defined as at least chronic moderate symptoms which frequently interfere with daily activities and require anti-asthma/anti-inﬂammatory agents
* Have received immunomodulating agents (including immunosuppressive agents, interferon or other immune or cytokine-based therapies), immunisation, and/or systemic chemotherapeutic agents within 60 days of Screening or expected to receive these agents during the course of the study
* Recipient of live attenuated vaccines within 60 days of Screening
* Recipient of whole killed, toxoid or sub-unit vaccines (e.g. influenza, pneumococcus, tetanus, hepatitis B) within 42 days prior to Baseline
* Ever received an HIV prophylactic or immunotherapeutic vaccine (does not apply to subjects who have written documentation of receiving placebo or adjuvant only)
* Recreational and/or therapeutic drug or alcohol use that, in the opinion of the Investigator, might compromise the subject's participation in any way.
* Medical or psychiatric condition or occupational responsibilities that may preclude compliance with the protocol
* Laboratory blood values:

  * Haemoglobin <11.0 grams/decilitre (g/dL) for men and <10.0 g/dL for women
  * Neutrophil count <800/mm3
  * Platelet count <50,000/mm3
  * Aspartate aminotransferase or Alanine transaminase >2.5 times Upper Limit of Normal (ULN)
  * Lipase >2.5 times ULN
  * Amylase >1.5 times ULN (unless serum lipase is ≤1.5 times ULN)
  * Subjects with an estimated creatinine clearance of <80 mL/minute
* Recipients of blood products or immunoglobulins within 6 months prior to Screening or loss of 450 mL or more of blood during the three months prior to Screening
* Recipients of experimental or investigational agents within 30 days prior to Screening
* Previous participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety | Several points throughout the 12 week active phase and 12 week and follow up period
  Examined through treatment-emergent adverse events, vital signs and routine laboratory screening.

SECONDARY OUTCOMES:
Immunogenicity | Several points throughout the 12 week active phase and 12 week and follow up period
  Immunogenicity will be assessed by ELISpot and other markers of immune response
Impact on HIV infection | Several points throughout the 12 week active phase and 12 week and follow up period
  Assessed by HIV-1 viral load and CD4 T-cell counts.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Kloverpris HN, Jackson A, Handley A, Hayes P, Gilmour J, Riddell L, Chen F, Atkins M, Boffito M, Walker BD, Ackland J, Sullivan M, Goulder P. Non-immunogenicity of overlapping gag peptides pulsed on autologous cells after vaccination of HIV infected individuals. PLoS One. 2013 Oct 4;8(10):e74389. doi: 10.1371/journal.pone.0074389. eCollection 2013. PMID 24124451
- [Derived] Jackson A, Kloverpris HN, Boffito M, Handley A, Atkins M, Hayes P, Gilmour J, Riddel L, Chen F, Bailey-Tippets M, Walker B, Ackland J, Sullivan M, Goulder P. A randomised, placebo-controlled, first-in-human study of a novel clade C therapeutic peptide vaccine administered ex vivo to autologous white blood cells in HIV infected individuals. PLoS One. 2013 Sep 17;8(9):e73765. doi: 10.1371/journal.pone.0073765. eCollection 2013. PMID 24069230